CLINICAL TRIAL: NCT06763939
Title: A Randomized, Comparative, Investigator-blinded Study to Evaluate the Efficacy of a Dermocosmetic Product RT00401 - Formula: GO0046 on Atopic Dermititis Severity in Subjects With Mild Atopic Dermatitis Versus Placebo.
Brief Title: Evaluation of the Efficacy of a Dermocosmetic Product RT00401-GO0046 on Atopic Dermititis Severity in Subjects With Mild Atopic Dermatitis Versus Placebo
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: RT0040120240799
Record Dates: First submitted 2024-12-20; First posted 2025-01-08 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Swab samplings on skin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects with mild atopic dermatitis: This is an intra-individual study. The included subjects will apply both products, one on each side of target areas. The target areas can be located on both arms, both legs, both feet, both sides of lower back, or both sides of face (for women only) or lower back if the zones are clearly distinct and accessible for the products application.
  One of the identified areas will be tested with RT00401-GO0046 cream and the symmetric area will be tested with RT00401-GA0677 cream according to randomization.
  Not all study participants will apply the products to the same sides.
  Interventions: Other: RT00401-GO0046; Other: RT00401-GA0677

INTERVENTIONS:
Other: RT00401-GO0046 — Cosmetic care product
Other: RT00401-GA0677 — Placebo cosmetic care product

SUMMARY:
The aim of this study is to evaluate the RT00401- GO0046 formula on atopic dermititis severity in subjects with mild atopic dermatitis versus placebo on 26 subjects.

The objectives of this study are:

* To evaluate the clinical efficacy of the RT00401-GO0046 cream compared to RT00401-GA0677 placebo cream on AD severity of tested areas and flare-up onset.
* To evaluate the effect of the RT00401-GO0046 cream on microbiota diversity and other pharmaco-clinical biomarkers with respective techniques on skin surface in subjects with AD compared to the effect of the RT00401-GA0677 placebo cream.
* To illustrate the effect of the RT00401-GO0046 cream with photos of the tested areas.

This study will be conducted as an intra-individual, comparative, randomized, monocentric, investigator-blinded study, with 3 visits are planned:

* Visit 1 (D1): Inclusion and 1st products application
* Visit 2 (D29 +/- 2 days): 1-month follow-up visit
* Visit X (Suspected flare-up +/- 2 days): End-of-study visit if AD flare-up is confirmed
* Visit 3 (D85 +/- 3 days): End-of-study visit This clinical study is designed as an investigator-blinded study. Participants will be required to apply two different products, one on each side: Product A and Product B. One of these products is the "test product" RT00401 Formula GO0646, and the other is the "control product" RT00401 Formula GA0677. However, participants will not know which product is which. The randomization will determine the side on which each product is applied (Product A on the right and Product B on the left, or vice versa). The product tubes will be identical, ensuring that neither the participants nor the investigator will know which product is the test product or the control product. This blinding ensures that neither the participants nor the investigator will be influenced by the nature of the products applied, thereby enhancing the robustness and objectivity of the study results.

ELIGIBILITY:
Main Inclusion criteria :

* Female and/or male;
* Subject aged ≥ 18 years;
* Subjects presenting atopic dermatitis according to the definition of "the U.K Working Party's Diagnostic Criteria for Atopic Dermatitis";
* Subject presenting a mild AD with a SCORAD from 15 to 20 with dryness evaluation parameter ≥ 2 at inclusion;
* Based on the subject's statements regarding their skin condition history:
* Subject with AD symmetric lesions, size from 10 to 15 cm² on both target areas;
* Subject who will likely present a flare-up during their participation according to investigator's opinion;

Main Non inclusion criteria

* Subject whose skin condition in the potential target areas is contact eczema or dyshidrotic eczema rather than atopic dermatitis (particularly on feet).
* Subject having any other dermatologic condition than Atopic Dermatitis, or characteristics (like tattoo) on the tested areas, liable to interfere with the study assessments according to investigator opinion;
* Subject having significant hair growth on tested areas;
* Subject presenting a flare-up at time of inclusion visit requiring a therapeutic care;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the investigation centre's panel. They will be selected on the basis of inclusion and non-inclusion criteria specific to the study and on their ability to comply with the constraints required by the protocol. They will be definitely included in the study after a specific interview and a clinical examination.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Evaluation of SCORAD | At baseline (Day 1) and at the final visit (Day 85 or Day X if the flare-up of AD is confirmed before Day 85),
  an examination of the face and body of the subject is carried out by the dermatologist in charge of the study to evaluate the initial intensity of atopic dermatitis by determination of SCORAD index
Evaluation of L-SCORAD | At baseline (Day 1), at Visit 2 (Day 29) and at the final visit (Day 85 or Day X if the flare-up of AD is confirmed before Day 85),
  The Local SCORAD is the evaluation of the objective parameters of the SCORAD will be assessed independently on both target areas by the Investigator
Evaluation of L-PO SCORAD | At baseline (Day 1), at Visit 2 (Day 29) and at the final visit (Day 85 or Day X if the flare-up of AD is confirmed before Day 85),
  The Local PO SCORAD will be evaluated by the subjects independently on the same target areas that L-SCORAD
Evolution of pruritus sensations using numerical rating scale (NRS) | At baseline (Day 1), at Visit 2 (Day 29) and at the final visit (Day 85 or Day X if the flare-up of AD is confirmed before Day 85),
  The subject will realize auto-scoring of pruritus independently on both target areas perceived (with average intensity over the last 3 days) using a Numeric Rating Scale from 0 (no pruritus) to 10 (severe discomfort sensations).
Microbiota diversity | At baseline (Day 1), at Visit 2 (Day 29) and at the final visit (Day 85 or Day X if the flare-up of AD is confirmed before Day 85),
  A total of 18 cutaneous samples per subject: 3 by cotton-swab samples per sampling area per time point will be taken at each study visit, on the study areas (identified at inclusion visit), will be carried out for analyses
Metabolomic features | At baseline (Day 1), at Visit 2 (Day 29) and at the final visit (Day 85 or Day X if the flare-up of AD is confirmed before Day 85),
  A total of 18 cutaneous samples per subject: 3 by cotton-swab samples per sampling area per time point will be taken at each study visit, on the study areas (identified at inclusion visit), will be carried out for analyses
Cytokine panel | At baseline (Day 1), at Visit 2 (Day 29) and at the final visit (Day 85 or Day X if the flare-up of AD is confirmed before Day 85),
  A total of 18 cutaneous samples per subject: 3 by cotton-swab samples per sampling area per time point will be taken at each study visit, on the study areas (identified at inclusion visit), will be carried out for analyses
Transepidermal water loss measurments by tewameter® | At baseline (Day 1), at Visit 2 (Day 29) and at the final visit (Day 85 or Day X if the flare-up of AD is confirmed before Day 85),
  A trans-epidermal water loss will be measured with a Tewameter TM 300® independently on both target areas
Skin pH measurements by phmeter | At baseline (Day 1), at Visit 2 (Day 29) and at the final visit (Day 85 or Day X if the flare-up of AD is confirmed before Day 85),
  A cutaneous pH level will be measured with a COURAGE & KHAZAKA PH 900 PC Skin pHmeter® fitted with an Ingold® electrode independently on both target areas
Investigator Global Assessment (IGA) | At baseline (Day 1), at Visit 2 (Day 29) and at the final visit (Day 85 or Day X if the flare-up of AD is confirmed before Day 85),
  IGA will be assessed by the investigator independently on both target areas perceived at each study visit from Visit 2, compared to Visit 1, according to a 5-point scale: 0= worse, 1= no change, 2= slight improvement, 3= marked improvement; 4= total resolution Local IGA assesses the evolution of target areas AD basing on objective signs (erythema, oedema/papulation, oozing/crusts, excoriation, lichenification, dryness) compared to baseline (Visit 1).
Patient Global Assessment (PGA) | At baseline (Day 1), at Visit 2 (Day 29) and at the final visit (Day 85 or Day X if the flare-up of AD is confirmed before Day 85),
  PGA will be assessed by the subjects independently on both target areas perceived at each study visit from Visit 2, compared to Visit 1, according to a 5-point scale: 0= worse 1= no change, 2= slight improvement, 3= marked improvement; 4= total resolution Local PGA assesses the evolution of target areas AD intensity compared to baseline (Visit 1).
Atopic dermititis severity by counting of flare-up onset | At the end of study, after last patient out, approximately 6 months after the beggining of the study.
  At the end of the study, the number of flare-ups that occurred during the study will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Dermscan Poland, Gdansk, Poland, Poland

IPD SHARING:
Plan to Share IPD: No